CLINICAL TRIAL: NCT02445846
Title: Field Performance Evaluation of Dual Rapid HIV & Syphilis Tests in Zambia
Brief Title: Dual Rapid HIV & Syphilis Tests in Zambia
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0528
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-02

CONDITIONS: HIV; Syphilis
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women, regardless of HIV status, seeking antenatal care at clinics in Lusaka, Zambia
  Interventions: Device: dual HIV/syphilis rapid diagnostics tests

INTERVENTIONS:
Device: dual HIV/syphilis rapid diagnostics tests
  Other Names: Chembio and Standard Disgnostics

SUMMARY:
The purpose of this study is to provide evidence on the performance and operational characteristics of commercially available dual HIV/syphilis Rapid Diagnostic Tests (RDTs) in Zambia for their introduction into antenatal care and other settings.

DETAILED DESCRIPTION:
Early detection and timely intervention of pregnant women infected with HIV and/or syphilis is critical. To improve the number of women tested and treated, the Centre for Infectious Disease Research in Zambia (CIDRZ) and the Ministry of Community Development, Mother and Health (MCDMCH) this field study will assess the effectiveness of newly developed dual HIV and syphilis rapid diagnostic tests (RDTs) manufactured by Chembio and Standard Diagnostics in Lusaka District antenatal clinics.

The specific objectives of this field performance evaluation of the rapid diagnostics are to determine the antenatal clinic-based performance of dual HIV/syphilis RDTs compared to that of current reference standard assays, and to assess the operational characteristics and acceptability of these dual HIV/syphilis RDTs to patients and health care providers This cross-sectional study of 3,765 pregnant women will validate the performance of Chembio and Standard Diagnostics dual HIV and Syphilis RDTs.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending their first antenatal care visit at a study clinic
* 18 years of age or older
* Willing and able to provide informed consent for study participation

Exclusion Criteria:

* Prior participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women, regardless of HIV status, seeking antenatal care at Chipata, Chawama, or Kamwala District Health Centres in Lusaka, Zambia.
Sampling Method: Non-Probability Sample
Enrollment: 3010 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
performance of dual rapid HIV/syphilis tests | day 1/enrollment
  The performance of the rapid study tests will be assessed by determining the specificity and the sensitivity when compared to reference standard assays

SECONDARY OUTCOMES:
acceptability of use of dual rapid HIV/syphilis tests | day 1/enrollment
  the operational characteristics and acceptability of the tests to patients and health care providers will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kasaro, MBChB, MSc, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Katepa-Bwalya M, Kankasa C, Babaniyi O, Siziya S. Effect of using HIV and infant feeding counselling cards on the quality of counselling provided to HIV positive mothers: a cluster randomized controlled trial. Int Breastfeed J. 2011 Sep 26;6:13. doi: 10.1186/1746-4358-6-13. PMID 21943308
- [Background] Kalichman SC, Pellowski J, Turner C. Prevalence of sexually transmitted co-infections in people living with HIV/AIDS: systematic review with implications for using HIV treatments for prevention. Sex Transm Infect. 2011 Apr;87(3):183-90. doi: 10.1136/sti.2010.047514. Epub 2011 Feb 17. PMID 21330572
- [Background] Lee MJ, Hallmark RJ, Frenkel LM, Del Priore G. Maternal syphilis and vertical perinatal transmission of human immunodeficiency virus type-1 infection. Int J Gynaecol Obstet. 1998 Dec;63(3):247-52. doi: 10.1016/s0020-7292(98)00165-9. PMID 9989893
- [Background] Mwapasa V, Rogerson SJ, Kwiek JJ, Wilson PE, Milner D, Molyneux ME, Kamwendo DD, Tadesse E, Chaluluka E, Meshnick SR. Maternal syphilis infection is associated with increased risk of mother-to-child transmission of HIV in Malawi. AIDS. 2006 Sep 11;20(14):1869-77. doi: 10.1097/01.aids.0000244206.41500.27. PMID 16954728
- [Background] WHO. Progress Report 2010; Towards Universal Access: Scaling up priority HIV/AIDS interventions in the health sector; Chapter 5: Scaling Up HIV Services for Women and Children http://www.who.int/hiv/pub/2010progressreport/ch5_en.pdf. Accessed July 12, 2011.
- [Background] Watson-Jones D, Changalucha J, Gumodoka B, Weiss H, Rusizoka M, Ndeki L, Whitehouse A, Balira R, Todd J, Ngeleja D, Ross D, Buve A, Hayes R, Mabey D. Syphilis in pregnancy in Tanzania. I. Impact of maternal syphilis on outcome of pregnancy. J Infect Dis. 2002 Oct 1;186(7):940-7. doi: 10.1086/342952. Epub 2002 Sep 3. PMID 12232834
- [Background] Watson-Jones D, Gumodoka B, Weiss H, Changalucha J, Todd J, Mugeye K, Buve A, Kanga Z, Ndeki L, Rusizoka M, Ross D, Marealle J, Balira R, Mabey D, Hayes R. Syphilis in pregnancy in Tanzania. II. The effectiveness of antenatal syphilis screening and single-dose benzathine penicillin treatment for the prevention of adverse pregnancy outcomes. J Infect Dis. 2002 Oct 1;186(7):948-57. doi: 10.1086/342951. Epub 2002 Sep 3. PMID 12232835
- [Background] Gerbase AC, Rowley JT, Heymann DH, Berkley SF, Piot P. Global prevalence and incidence estimates of selected curable STDs. Sex Transm Infect. 1998 Jun;74 Suppl 1:S12-6. PMID 10023347
- [Background] McDermott J, Steketee R, Larsen S, Wirima J. Syphilis-associated perinatal and infant mortality in rural Malawi. Bull World Health Organ. 1993;71(6):773-80. PMID 8313495
- [Background] Di Mario S, Say L, Lincetto O. Risk factors for stillbirth in developing countries: a systematic review of the literature. Sex Transm Dis. 2007 Jul;34(7 Suppl):S11-21. doi: 10.1097/01.olq.0000258130.07476.e3. PMID 17592385
- [Background] Strasser S, Bitarakwate E, Gill M, Hoffman HJ, Musana O, Phiri A, Shelley KD, Sripipatana T, Ncube AT, Chintu N. Introduction of rapid syphilis testing within prevention of mother-to-child transmission of HIV programs in Uganda and Zambia: a field acceptability and feasibility study. J Acquir Immune Defic Syndr. 2012 Nov 1;61(3):e40-6. doi: 10.1097/QAI.0b013e318267bc94. PMID 22820810
- [Background] Kettler H, White K, Hawkes S. Mapping the landscape of diagnostics for sexually transmitted infections. World Health Organization, Geneva, 2004.